CLINICAL TRIAL: NCT06572800
Title: Use of DiviTum-TKa as a Biomarker Assay for CDK4/6 Inhibitor Medication Compliance and Drug-Drug Interaction Assessment in ER/PR Positive Metastatic Breast Cancer
Brief Title: Tka Assay for CDK4/6i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000033797; NCI-2024-01395 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000033797 (Other: Yale University); P30CA016359 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic HER2-Negative Breast Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Health services research (DiviTum-TKa) (Experimental): Patients undergo collection of blood samples per SOC on days 1, 15, and 28 of cycle 1, days 15 and 28 of cycle 2, days 15 and 28 of cycle 3, and day 28 of subsequent cycles for up to 12 cycles for analysis by DiviTum-TKa in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: DiviTum-TKa

INTERVENTIONS:
Device: DiviTum-TKa — Analyze blood samples by DiviTum-TKa

SUMMARY:
This clinical trial assesses whether using a test developed by DiviTum can identify optimal levels of CDK 4/6 inhibitor medications in the blood and whether assessing medical compliance and drug-drug interactions can optimize (improve) these levels in patients with estrogen receptor (ER) or progesterone receptor (PR) positive, and human epidermal growth factor receptor 2 (HER2)-negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and are receiving CDK 4/6 inhibitors. CDK4/6 inhibitors in combination with endocrine therapy (ET) is first line treatment for metastatic hormone positive (ER/PR positive) breast cancer (mBC). Thymidine kinase is a biomarker (biological molecule found in blood, other body fluids, or tissues that is a sign of a condition or disease) that reflects cell proliferation (an increase in the number of cells as a result of cell growth and cell division). DiviTum-thymidine kinase activity (TKa) is a Food and Drug Administration approved assay which showed that a TKa is associated with the decreased likelihood of disease progression within 30 days or 60 days post testing. Using the DiviTum-TKa may improve medication compliance and remove potential drug-drug interactions in patients with ER/PR positive HER2-negative MBC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the rate of improvement in CDK4/6 inhibitor response (i.e. moving from profile 3 to profiles 1 or 2) in cycles 2 and 3 after counseling for medication compliance and adjustment of potential deleterious drug-drug interactions.

SECONDARY OBJECTIVES:

I. Estimate the rate of sub-optimal CDK 4/6 inhibitor response (profile 3) in patients with metastatic hormone positive breast cancer in cycle 1 of CDK4/6 inhibitor and endocrine therapy in the first line setting.

II. Compare clinical benefit rate (CBR) in patients with sub-optimal (profile 3) and optimal (profiles 1 and 2) CDK4/6 inhibitor response after both cycles 1 and cycle 3.

III. Compare progression free survival (PFS) rates at 6 months (mo), 12 mo, 18 mo in patients with sub-optimal (profile 3) and optimal (profiles 1 and 2) CDK 4/6 inhibitor response after both cycles 1 and cycle 3.

IV. Assess CDK4/6 inhibitor response via TKa levels upon CDK4/6 inhibitor dose reductions or changes in CDK4/6 inhibitor regimens.

V. Compare CDK4/6 inhibitor response profiles across the three CDK 4/6 inhibitors among different patients and within the same patients if CDK4/6 inhibitor is changed throughout treatment course.

VI. Correlate TKa levels with tumor marker levels. VII. Assess plasma concentrations of CDK4/6 inhibitor drugs in patients with suboptimal TKa levels.

OUTLINE:

Patients undergo collection of blood samples per standard of care (SOC) on days 1, 15, and 28 of cycle 1, days 15 and 28 of cycle 2, days 15 and 28 of cycle 3, and day 28 of subsequent cycles for up to 12 cycles for analysis by DiviTum-TKa in the absence of disease progression or unacceptable toxicity.

After completion of study intervention, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed metastatic ER-positive (> 10%), PR-positive or PR-negative, and HER2-negative (0 by immunohistochemistry [IHC] or if +1 or +2 by IHC, not amplified by fluorescence in situ hybridization [FISH]) breast cancer; ER positivity, PR positivity, and HER2 negativity as per the 2018 joint American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Participants must be starting CDK4/6 inhibitor and endocrine therapy as part of first-line therapy per standard of care and be previously CDK4/6 inhibitor-naïve.
* Participants must be enrolled prior to starting CDK4/6 inhibitor therapy.
* Participants must be ≥ 18 years of age.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status < 3.
* Willing and able to provide written informed consent for the trial.

Exclusion Criteria:

* Participants without evidence of metastatic disease prior to registration.
* Participants with prior use of CDK4/6 inhibitor therapy.
* Participants who are unable to provide informed consent for the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with thymidine kinase activity (TKa) values that switch from profile 3 to profile 1 or 2 after medication compliance and drug-drug interaction assessment | Immediately following counseling for medication compliance and adjustment of potential deleterious drug-drug interactions
  Will be estimated using the two-sided 95% exact confidence interval (CI) using Clopper-Pearson method.
Rate of improvement in CDK4/6 inhibitor response (i.e. moving from profile 3 to profiles 1 or 2) | At day 28 of cycles 2 and 3 immediately following counselling for medication compliance and removing potential deleterious drug-drug interactions
  Will be estimated using the two-sided 95% exact CI using Clopper-Pearson method.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) in patients with sub-optimal (profile 3) and optimal (profiles 1 and 2) CDK4/6 inhibitor response | At day 28 of cycles 1 and 3
  CBR is defined as the total number of patients who achieve a complete response, partial response, or stable disease for 6 months or more from day 1 (D1) cycle 1 (C1). Comparisons between paired outcomes will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest.
Progression free survival (PFS) | At 6, 12, and 18 months
  PFS is defined as the time from D1C1 to disease progression. Will be estimated using Kaplan-Meier method.
CDK4/6 inhibitor response via TKa levels upon CDK4/6 inhibitor dose reductions or changes in CDK4/6 inhibitor regimen due to adverse events | Up to 2 years
  Will estimate the two-sided 95% exact CI using Clopper-Pearson method.
Comparison of CDK4/6 inhibitor response profiles across the three CDK 4/6 inhibitors | Up to 2 years
  Will be completed using the paired t-test or Wilcoxon signed-rank test for continuous parameters of interest, or McNemar's Chi-square test for categorical parameters of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Rozenblit, Principal Investigator — Yale University
Locations (18):
- United States (18):
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island

IPD SHARING:
Plan to Share IPD: No